CLINICAL TRIAL: NCT04831255
Title: A Stratified Investigation of a Single Injection of ZILRETTA™ (Triamcinolone Acetonide Extended-release Injectable Suspension) for Symptomatic Relief in Patients With Idiopathic Adhesive Capsulitis of the Shoulder
Brief Title: ZILRETTA™ for Treatment of Idiopathic Adhesive Capsulitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not able to find enough subjects
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Brian Werner, MD, Assistant Professor, Department of Orthopaedic Surgery, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21584
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder; Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: All subjects receive the ZILRETTA injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ZILRETTA (Experimental): Single injection of triamcinolone acetonide extended-release injectable suspension, injected in the glenohumeral joint under ultrasound guidance.
  Interventions: Drug: triamcinolone acetonide extended-release injectable suspension

INTERVENTIONS:
Drug: triamcinolone acetonide extended-release injectable suspension — ZILRETTA (triamcinolone acetonide extended-release injectable suspension) injection in the glenohumeral joint administered under ultrasound guidance.
  Other Names: ZILRETTA

SUMMARY:
Adhesive capsulitis is a fairly common orthopedic condition that causes pain and loss of range of motion. There are a variety of ways to treat adhesive capsulitis, one of them being an intra-articular steroid injection. This is done to help decrease the inflammatory response caused by adhesive capsulitis. In this study, all participants will receive an intra-articular glenohumeral injection of ZILRETTA and will be followed up with at four time points over 1 year to observe pain, function and range of motion following the injection.

DETAILED DESCRIPTION:
Adhesive capsulitis is a painful shoulder condition characterized by a gradual loss of both passive and active range of motion due to inflammatory changes and eventual fibrosis and contracture of the shoulder joint capsule. It occurs in about 2% to 5% of the population, and a majority of patients are female. The true cause of the condition remains unclear, however, it has been proposed that the initial synovitis stimulates the development of a fibrotic cascade. The development of adhesive capsulitis has been associated with diabetes mellitus, thyroid dysfunction, Dupuytrens contractures, autoimmune diseases and treatments for certain cancers. Adhesive capsulitis progresses through four predictable phases, defined by symptoms, physical examination, arthroscopic appearance and biopsies.

Regardless of stage, the mainstay of treatment for adhesive capsulitis of the shoulder is conservative, focused mainly on physical therapy combined with a home exercise program, regardless of stage. Pharmacologic agents are often used as adjuncts to physical therapy, and include nonsteroidal anti-inflammatory medications (NSAIDs), oral corticosteroids and intra-articular injections of corticosteroids. Although a large percentage of patients in the early stages of disease respond well to conservative treatments, those who fail therapy and injections may require surgical intervention, including arthroscopy with lysis of adhesions and/or manipulation under anesthesia.

Numerous studies have investigated the effect and success of injections combined with standard physical therapy for adhesive capsulitis of the shoulder. In general, intra-articular injection of corticosteroids has been found to be superior to administration of oral cortisone and at least equivalent to manipulation under anesthesia alone. Injections have been shown to reduce pain quicker and result in earlier return of range of motion. Low doses of steroid appear equally as effective as higher doses. Image-guided injections, whether ultrasound or fluoroscopic guided injections, have also been shown to be more effective than blinded injections.

Failure of an injection and therapy to provide relief either results in a repeat image-guided injection or surgical intervention, both of which have significant associated cost and potential morbidity. Thus, there would be significant potential value to a long-acting, sustained release intra-articular steroid injection for the treatment of adhesive capsulitis of the shoulder. Zilretta®, triamcinolone acetonide extended release suspension 32 mg, is a microsphere formulation of injectable steroid which is FDA-approved for and has shown significant promise for the treatment of knee osteoarthritis. This long-acting steroid could have several important advantages in the treatment of shoulder adhesive capsulitis. It may potentiate and prolong the anti-inflammatory effect of the steroid, and potentially avoid the need for costly additional image-guided injections or expensive and potentially morbid surgery. An additional potential benefit is less elevation of peripheral blood glucose in diabetics, a known complication of traditional steroid injections that has been demonstrated to be mitigated using a sustained release formulation.

Out primary aim in this study is to assess patient reported pain and outcomes in patients with idiopathic adhesive capsulitis of the shoulder at 3, 6 and 12 months following single, image guided ZILRETTA injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic adhesive capsulitis (onset <6 months prior)
* Pain rating of 5 or greater out of 10 on 0-10 scale at time of enrollment
* Willing to come on site for follow up evaluations at 1 month, 3 months, 6 months, and 12 months after the injection

Exclusion Criteria:

* Active workers compensation case
* Known psychiatric disorders under active treatment
* Uncontrolled diabetes (defined as diabetic ketoacidosis, severe peripheral neuropathy, ophthalmologic or renal manifestations)
* Diagnosed osteoarthritis of the ipsilateral or contralateral shoulder
* Painful joint condition in another part of the body affecting perceived pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Score | 6 months after injection
  Pain rating on a scale of 0-10, higher numbers indicating a worse outcome

SECONDARY OUTCOMES:
American Shoulder and Elbow Society Score | 6 months after injection
  Pain and function patient reported outcome for the shoulder. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
American Shoulder and Elbow Society Score | 12 months after injection
  Pain and function patient reported outcome for the shoulder. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
PROMIS Physical Function Score | 6 months after injection
  Patient reported outcome measuring physical function level measured by T scores and standard deviations. The average is 50, so a T score lower than 50 indicates a worse outcome.
PROMIS Physical Function Score | 12 months after injection
  Patient reported outcome measuring physical function level measured by T scores and standard deviations. The average is 50, so a T score lower than 50 indicates a worse outcome.
Triplanar Range of Motion | 1 month after injection
  Shoulder range of motion
Triplanar Range of Motion | 3 months after injection
  Shoulder range of motion
Triplanar Range of Motion | 6 months after injection
  Shoulder range of motion
Triplanar Range of Motion | 12 months after injection
  Shoulder range of motion
Need for another injection | 12 months after injection
  Yes or no answer if the patient needed another corticosteroid injection during their time enrolled in the study
Time to second injection (if applicable) | 12 months after injection
  how long after the ZILRETTA injection the patient needed another corticosteroid injection

CONTACTS AND LOCATIONS:
Overall Officials: Brian Werner, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT04831255/ICF_000.pdf